CLINICAL TRIAL: NCT03780062
Title: Interest of S100B Protein for Patient Victim of Minor Traumatic Brain Injury and Treated by Antiplatelet
Acronym: PETEChIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETEChIA
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Minor Traumatic Brain Injury; Treatment by Antiplatelet
Keywords: S100B protein; minor traumatic brain injuries; antiplatelet therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S100B protein dosing (Experimental)
  Interventions: Biological: S100B protein dosing

INTERVENTIONS:
Biological: S100B protein dosing — Patients under antiplatelet therapy and who have a minor traumatic brain injury will have a blood samples with protein S100B dosage on arrival to the emergency room and after they will have a brain scanner between 4 and 8 hours after the trauma to analyse the negative predictive value with a treshold of 0.105 μg/L

SUMMARY:
All the patients admitted in emergency department for minor traumatized cranial, with antiplatelet therapy, can be included, after checked inclusion and non inclusions criterias. If they are agree, a blood sample for the dosage of S100b will be done.

No other modification of the medical care, all patients will have tomodensitometria, according with recommendations. The aim of the study is to validate the negative predictive value of S100b in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Years old
* Minor traumatic brain injury measured by a Glasgow score between 13 and 15
* Antiplatelet agent therapy
* Free subject without tutorship or curatorship

Exclusion Criteria:

* Age < 18 years old
* Glasgow score <13
* Traumatic brain injury older than 6 hours
* Patient without any social security system
* Patient with renforced protection (tutorship, curatorship, …)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Brain scanner Detection of a cerebral lesion requiring a surgery or medical intervention or an hospitalisation for a patient who have serum level of S100B protein with the treshold of 0.105 μg/L | 3 hours

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU of MONTPELLIER, Montpellier
  - CHU of NICE, Nice
  - La Pité Salpêtrière, Paris
  - CHU of POITIERS, Poitiers